CLINICAL TRIAL: NCT03020849
Title: Can we Define a Clinical Score for Predicting of Hypofibrinogenemia in Severe Trauma
Brief Title: Predictors of Hypofibrinogenemia in Severe Trauma
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0015
Record Dates: First submitted 2017-01-10; First posted 2017-01-13 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-01

CONDITIONS: Severe Trauma
Keywords: hypofibrinogenemia; prediction score; severe trauma
MeSH Terms: conditions — Wounds and Injuries; Afibrinogenemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this retrospective and prospective study, the aim is to determine a score for predicting a fibrinogen <1.5g/L (corresponding to European threshold of Directors recommendations of fibrinogen concentrates)

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* severe trauma

Exclusion Criteria:

* age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe trauma
Sampling Method: Non-Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
rate of fibrinogen in blood sample at hospitalisation | day 0 (at hospitalisation)
  This fibrinogen rate is correlated to pre-hospital and admission clinical parameters (trauma type, physiologic status, treatments administered, biologic checkup) to predict fibrinogenemia at hospitalisation

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - HEH - Hospices Civils de Lyon, Lyon
  - CHLS, Hospices Civils de Lyon, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No